CLINICAL TRIAL: NCT07392996
Title: Does Early Postoperative Fluid Management Affect Functional Delayed Graft Function After Living Donor Kidney Transplantation? A Retrospective Cohort Analysis
Brief Title: Does Early Postoperative Fluid Management Affect Functional Delayed Graft Function After Living Donor Kidney Transplantation?
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hatice Güneş Yeşilova, MD, Principal Investigator, Ankara University
Other Study IDs: RENALTRANSAÜTF
Record Dates: First submitted 2026-01-16; First posted 2026-02-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Renal Transplant; DGF
Keywords: Kidney transplantation; fDGF; fluid replacement; living organ donor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fluid management in renal transplantation is of critical importance for optimizing graft function and minimizing complications such as delayed graft function (DGF) and acute kidney injury (AKI). The aim of this study was to retrospectively investigate the effects of early postoperative (the first 4 hours after transplantation) fluid replacement volume on graft function in patients undergoing living donor kidney transplantation.

DETAILED DESCRIPTION:
Maintaining an appropriate fluid balance is of paramount importance in renal transplantation. Overhydration may lead to complications such as pulmonary edema and impaired renal perfusion, whereas insufficient hydration can result in hypoperfusion and acute kidney injury (AKI). The amount of fluid administered in conjunction with goal-directed hemodynamic management plays a crucial role in improving kidney transplant outcomes. By carefully balancing fluid therapy and monitoring hemodynamic parameters, graft function can be improved and postoperative complications can be reduced.

Delayed graft function (DGF) is a term used instead of post-transplant acute renal failure and is broadly defined as the need for dialysis within the first week after transplantation. It is well known that DGF increases susceptibility to acute rejection. Implementing interventions before irreversible injury occurs represents the most effective strategy for reducing DGF. Fluid therapy has been shown to be effective in preventing AKI in selected patient populations.

Several factors predispose kidney transplant recipients to hypotension, including the sudden redistribution of approximately 25% of the cardiac output to the renal graft following revascularization, the release of vasoactive mediators accumulated during ischemia with the associated risk of post-reperfusion syndrome, and cytokine-mediated hypotension related to immunosuppressive agents administered shortly before vascular unclamping. In addition, the transplanted kidney is denervated and lacks neurogenic regulation of renal blood flow. Consequently, renal perfusion becomes more dependent on intravascular volume status and arterial blood pressure. Every effort should therefore be made to maintain adequate arterial blood pressure, primarily through sufficient intravascular volume and secondarily through the judicious use of vasopressors when necessary.

Despite improvements in overall outcomes among kidney transplant recipients, delayed graft function remains a significant complication and an important predictor of subsequent clinical outcomes. DGF is associated with reduced graft and patient survival, long-term graft dysfunction, and an increased incidence of acute rejection. Optimized perioperative hemodynamic management has been shown to be effective in preventing DGF and reducing perioperative complications; however, the optimal strategy for fluid therapy remains controversial.

Kidney transplant recipients are at risk for developing DGF, AKI, and fluid overload. Hypovolemia may exacerbate renal injury, whereas excessive fluid administration may result in pulmonary edema.

Previous studies investigating optimal fluid replacement strategies have focused on targeting central venous pressure (CVP), restrictive fluid regimens or goal-directed fluid therapy, and the timing of fluid administration; however, no consistent conclusions have been reached.

One study evaluating the effects of a restrictive fluid regimen demonstrated an approximately fourfold increase in the risk of DGF. Another study showed that patients who received the largest volume of fluid immediately before renal artery unclamping exhibited lower hemodynamic instability and higher systolic blood pressure, mean arterial pressure, and central venous pressure levels. In contrast, a retrospective study examining goal-directed fluid replacement reported adverse effects on clinical outcomes ; however, these findings are inconsistent with other studies investigating goal-directed fluid therapy.

Optimizing fluid management in renal transplantation remains a critical component of improving patient outcomes and ensuring long-term graft success. In our clinical practice, we aim to investigate the effects of early postoperative fluid replacement volumes on graft function and patient outcomes, with the goal of contributing to improved clinical practices and better long-term outcomes for transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients and donors aged 18 years and older
* Renal transplant from a living donor

Exclusion Criteria:

* Patients under 18 years of age
* Patients with incomplete or missing medical records
* Patients with heart disease (ejection fraction < 30)
* Multiple organ transplant
* History of repeated kidney transplants
* Cadaveric renal transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between 2017 and 2025, 122 patients who met the inclusion criteria for the study were enrolled from among recipients and donors of living donor renal transplants performed in the General Surgery operating theatre at Ankara University İbni Sina Research and Application Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Functional Delayed Graft Function (fDGF) | postoperatif 7 days
  Functional delayed graft function (fDGF) was defined as the absence of a spontaneous daily decrease of at least 10% in serum creatinine levels for three consecutive days during the first postoperative week. To avoid misclassification in patients with excellent early graft function, a lack of creatinine decline on postoperative day 3 was not classified as fDGF if optimal graft function had already been achieved by postoperative day 2.

SECONDARY OUTCOMES:
Kidney transplant function | Postoperative 1 year
  Graft dysfunction was defined as either the development of a need for hemodialysis or the presence of chronic allograft dysfunction, both occurring within the first postoperative year.
  Chronic allograft dysfunction (CKD-T) was defined as persistent graft dysfunction lasting for at least 3 months, characterized by an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m² and/or evidence of structural kidney damage in kidney transplant recipients.

CONTACTS AND LOCATIONS:
Overall Officials: Süheyla Karadağ Erkoç, Study Director — Ankara University İbni Sina Research and Application Hospital.
Locations (1):
- Ankara University İbni Sina Research and Application Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.